CLINICAL TRIAL: NCT04315090
Title: Post-surgical Outcomes Measure Using the ERAS Protocol for Posterior Cervical Decompression and Fusion
Status: Withdrawn | Type: Observational
Why Stopped: Personnel change and inadequate resources to proceed with the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew T. Neal, Principal Investigator, Mayo Clinic
Other Study IDs: 19-006598
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Degenerative Spinal Arthritis; Cervical Myelopathy; Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study is being conducted to help improve the pre-operative, intra-operative, and post-operative course for patients and enhance recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 89
* Diagnosis of cervical myelopathy, cervical stenosis, cervical disc disorder, or cervical spondylolisthesis

Exclusion Criteria:

* Cervical injury as the indication for surgery
* Emergent surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults scheduled to undergo posterior cervical spinal fusion.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-09 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | Will record length of stay in days 3 months following admission date.
  We will record the length of stay (date of admission to date of discharge) for the operative admission at the time of discharge.

SECONDARY OUTCOMES:
Rate of readmission | Within 3 months of discharge
Numerical rating scale (NRS)- pain | immediately before, immediately after, and 3 months after surgery
  Numerical score of neck pain. Scored 0 to 10. 10 is the worst pain.
SF-12 short form | immediately before, immediately after, and 3 months after surgery
  SF-12 short form health survey. Scored 0 to 100. 100 is the highest level of health.
Oswestry Disability Index | immediately before, immediately after, and 3 months after surgery
  questionnaire regarding low back pain. Scored 0 to 100. 100 being most severe disability.
Number of sessions with physical therapy and occupational therapy | will record number of physical and occupational therapy sessions during surgical admission 3 months following admission date
  record of number of sessions completed with physical or occupational therapy during the operative admission. We will determine this number at the time of discharge. We will calculate this number only once.
Disposition status | will record discharge disposition 3 months following surgical admission date
  We will determine the disposition status at the time of discharge following the operative admission. We will do this only once.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Neal, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials